CLINICAL TRIAL: NCT04313777
Title: The Evaluation of Virtual Reality Therapy Efficacy in the Treatment of Depressive and Anxiety Symptoms in Patients With Coronary Artery Disease
Brief Title: Virtual Reality Therapy in Cardiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wroclaw University of Health and Sport Sciences (Other)
Collaborators: Foundation for Senior Citizen Activation SIWY DYM (Other)
Responsible Party: Principal Investigator, Joanna Szczepańska-Gieracha, Professor, Wroclaw University of Health and Sport Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 59/0203/S/03
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Cardiovascular Diseases; Coronary Artery Disease; Depressive Symptoms; Mood Disorders; Anxiety; Stress
Keywords: virtual reality; cardiac rehabilitation; psychotherapy; cardiac surgery; depression; anxiety; stress
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Depression; Mood Disorders; Anxiety Disorders | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR therapy group (Experimental): Cardiac rehabilitation supplemented by VR therapy
  Interventions: Behavioral: Cardiac rehabilitation; Device: Virtual therapeutic support
- Control Group (Active Comparator): Cardiac rehabilitation supplemented by Schultz Autogenic Training
  Interventions: Behavioral: Cardiac rehabilitation; Behavioral: Schultz Autogenic Training

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — Four weeks of cardiac rehabilitation conducted in an outpatient care facility. Three times per week (80 minutes per day) cardiologically monitored aerobic training consisting of: 40 minutes of interval training on a cycloergometer and 40 minutes of general fitness exercises.
Device: Virtual therapeutic support — 8 sessions of VR therapy (each of them 20 minutes long). As a virtual reality source, VR Tier One device (Stolgraf®) were used. Thanks to using head mounted display and the phenomenon of total immersion VR therapy provides an intense visual, auditory and kinesthetic stimulation. It can have a calming and mood-improving effect or help the patients recognize their psychological resources and motivate to the rehabilitation process. In the virtual therapeutic garden there are a rich set of symbols and metaphors based on Ericksonian Psychotherapy approach.
  Arms: VR therapy group
Behavioral: Schultz Autogenic Training — 8 sessions of Schultz Autogenic Training (each of them 20 minutes long).
  Arms: Control Group

SUMMARY:
This study evaluates the effectiveness of virtual reality (VR) therapy in the treatment of depression and anxiety symptoms in patients undergoing second stage of cardiac rehabilitation. Half of the study group will receive VR therapy (VR group) as an addition to cardiologically monitored physical training. The other half of the group (control group) will receive Schultz Autogenic Training as a standard supplement to cardiological training

DETAILED DESCRIPTION:
Cardiologically monitored physical training in second stage of cardiac rehabilitation leads to the improvement in the physical capacity and overall fitness of the patients with cardiovascular diseases, allowing restoration of independence in daily functioning. Psychological support is required in order to reduce the negative psychological symptoms related to the heart disease. In this study the investigators want to assess the effectiveness of the virtual reality (VR) therapy compared to standard psychological support (Schultz Autogenic Training).Thanks to using head mounted display (VR goggles) and the phenomenon of total immersion VR therapy allows to completely separate the patient from the hospital environment, provides an intense visual, auditory and kinesthetic stimulation. Depending on the stage of therapy it can have a calming and mood-improving effect or, in another part of the therapy, it can motivate the patient to the rehabilitation process. The additional aim of the VR therapy is to help the patients regain their emotional balance, let them recognize their psychological resources and trigger the natural recovery mechanisms.

The aims of the project:

1. The evaluation of the influence of VR therapy on the depressive symptoms and the anxiety level of the patients undergoing second stage of cardiac rehabilitation.
2. The evaluation of the influence of VR therapy on the stress level of the patients undergoing second stage of cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Coronary Artery Disease;
* the second stage of cardiac rehabilitation conducted in outpatient settings;

Exclusion Criteria:

* cognitive impairment (MMSE<24);
* inability to self-complete the research questionnaires;
* presence of the following issues at the time of the examination or in the medical data: disturbances of consciousness, psychotic symptoms or other serious psychiatric disorders;
* initiation of psychiatric treatment during the research project;
* contraindications for virtual therapy (epilepsy, vertigo, eyesight impairment);
* the patient's refusal at any stage of the research project.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-04-03 (Actual)

PRIMARY OUTCOMES:
Change in depressed mood and anxiety from baseline | At baseline and after 8 sessions of VR therapy (week 3)
  The Hospital Anxiety and Depression Scale (HADS) is a fourteen-item scale scoring from 0 to 3 for each item. The first seven items relate to anxiety (HADS-A), and the remaining seven items relate to depression (HADS-D). The global scoring ranges from 0 to 42 with a cut-off point of 8/21 for anxiety and 8/21 for depression. The higher the score, the greater anxiety or depression symptoms. HADS will be performed at the beginning and after four weeks of treatment.

SECONDARY OUTCOMES:
Change in perception of stress from baseline | At baseline and after 8 sessions of VR therapy (week 3)
  The Perception of Stress Questionnaire (PSQ) is a 27-item scale scoring from 1 to 5 for each item. 21 items examine the level of stress in the area of emotional tension, external stress and intrapsychic stress, and 6 items refer to the lie scale. The global scoring for perception of stress ranges from 21 to 105 with a cut-off point of 60 for high level of perceived stress. The higher the score, the greater the sense of stress. PSQ will be performed at the beginning and after four weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Szczepańska-Gieracha, Prof., Principal Investigator — University School of Physical Education in Wroclaw, Poland; Sandra Jóźwik, MSc., Study Chair — University School of Physical Education in Wroclaw, Poland
Locations (2):
- Poland (2):
  - University School of Physical Education, Wroclaw, Lower Silesian Voivodeship
  - Centrum Kardiologiczne Pro Corde Sp. z o.o., Wroclaw, Lower Silesian Voivodeship

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Theng YL, Foo S. Game-based digital interventions for depression therapy: a systematic review and meta-analysis. Cyberpsychol Behav Soc Netw. 2014 Aug;17(8):519-27. doi: 10.1089/cyber.2013.0481. Epub 2014 May 8. PMID 24810933
- [Background] McCann RA, Armstrong CM, Skopp NA, Edwards-Stewart A, Smolenski DJ, June JD, Metzger-Abamukong M, Reger GM. Virtual reality exposure therapy for the treatment of anxiety disorders: an evaluation of research quality. J Anxiety Disord. 2014 Aug;28(6):625-31. doi: 10.1016/j.janxdis.2014.05.010. Epub 2014 Jun 7. PMID 25093964
- [Background] Maples-Keller JL, Bunnell BE, Kim SJ, Rothbaum BO. The Use of Virtual Reality Technology in the Treatment of Anxiety and Other Psychiatric Disorders. Harv Rev Psychiatry. 2017 May/Jun;25(3):103-113. doi: 10.1097/HRP.0000000000000138. PMID 28475502
- [Background] Freeman D, Reeve S, Robinson A, Ehlers A, Clark D, Spanlang B, Slater M. Virtual reality in the assessment, understanding, and treatment of mental health disorders. Psychol Med. 2017 Oct;47(14):2393-2400. doi: 10.1017/S003329171700040X. Epub 2017 Mar 22. PMID 28325167
- [Background] Valmaggia LR, Latif L, Kempton MJ, Rus-Calafell M. Virtual reality in the psychological treatment for mental health problems: An systematic review of recent evidence. Psychiatry Res. 2016 Feb 28;236:189-195. doi: 10.1016/j.psychres.2016.01.015. Epub 2016 Jan 12. PMID 26795129
- [Background] Szczepanska-Gieracha J, Morka J, Kowalska J, Kustrzycki W, Rymaszewska J. The role of depressive and anxiety symptoms in the evaluation of cardiac rehabilitation efficacy after coronary artery bypass grafting surgery. Eur J Cardiothorac Surg. 2012 Nov;42(5):e108-14. doi: 10.1093/ejcts/ezs463. Epub 2012 Aug 19. PMID 22906598
- [Background] Thompson T, Steffert T, Steed A, Gruzelier J. A randomized controlled trial of the effects of hypnosis with 3-D virtual reality animation on tiredness, mood, and salivary cortisol. Int J Clin Exp Hypn. 2011 Jan;59(1):122-42. doi: 10.1080/00207144.2011.522917. PMID 21104488
- [Derived] Dibben G, Faulkner J, Oldridge N, Rees K, Thompson DR, Zwisler AD, Taylor RS. Exercise-based cardiac rehabilitation for coronary heart disease. Cochrane Database Syst Rev. 2021 Nov 6;11(11):CD001800. doi: 10.1002/14651858.CD001800.pub4. PMID 34741536